CLINICAL TRIAL: NCT04571216
Title: Study Assessing Efficacy and Safety of NFL-101 as a Tobacco Cessation Therapy
Acronym: CESTO2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NFL Biosciences SAS (Industry)
Responsible Party: Principal Investigator, Yves Donazzolo, Principal Investigator, NFL Biosciences SAS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V10.1
Record Dates: First submitted 2020-09-15; First posted 2020-09-30 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Smoking Cessation; Nicotine Dependence
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Tobacco Products

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NFL-101 Dose 1 (Experimental): 50 µg per injection (in each arm), two injections at day 1, two injections at day 8, optional injections later on
  Interventions: Drug: NFL-101 dose 1
- NFL-101 Dose 2 (Experimental): 100 µg per injection (in each arm), two injections at day 1, two injections at day 8, optional injections later on
  Interventions: Drug: NFL-101 dose 2
- Placebo (Placebo Comparator): The placebo will consist of two syringes containing 1 mL of dilution solution, two injections at day 1, two injections at day 8, optional injections later on
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NFL-101 dose 1 — Subcutaneous injections
  Other Names: Tobacco leaf extract
  Arms: NFL-101 Dose 1
Drug: NFL-101 dose 2 — Subcutaneous injections
  Other Names: Tobacco leaf extract
  Arms: NFL-101 Dose 2
Drug: Placebo — Subcutaneous injections
  Other Names: WFI
  Arms: Placebo

SUMMARY:
CESTO 2 is a 318 participants, 3-arm, multicentric, randomized, double-blind, placebo-controlled Phase II clinical trial.

The main objectives are to select the most efficient dose and to assess long-term efficacy of NFL-101 compared to placebo, for abrupt cessation and for reduction before cessation.

DETAILED DESCRIPTION:
Long-term smoking cessation or reduction had been observed in thousands of patients when 1 or 2 subcutaneous injections of a desensitization treatment against tobacco allergy were taking place concomitantly with Target Quit Date (TQD). NFL Biosciences SAS developed a tobacco cessation drug candidate (NFL-101) consisting of a nicotine-free extract of tobacco proteins. According to the observations made during CESTO, a Phase I study on 24 smokers, NFL-101 appears to work by reducing cigarette appetence immediately and over a week after each injection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥ 18 and ≤ 70-year-old;
* With ECOG/WHO performance status 0-1 (Appendix 1);
* Subject currently smoking at least 11 cigarettes per day and with a dependency level ≥ 3 according to Fagerström Test for Nicotine Dependence scoring (see Appendix 2) [1];
* Subject willing to quit smoking;
* Good general health (i.e. no uncontrolled medical condition, or no medical condition that could interfere with the conduct and the outcomes of the study, according to the investigator);
* Good mental health (i.e. no alcohol or drug abuse in the past year, no psychiatric history- adequately treated depression is accepted);
* For women of childbearing potential: commitment to consistently and correctly use of a highly effective contraceptive measure: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner or sexual abstinence for the duration of the trial; (Females of non-childbearing potential: either surgically sterilized or at least 1 year postmenopausal (amenorrhoea duration at least 12 months)) ;
* Negative pregnancy test at screening visit;
* Laboratory parameters within the normal range of the laboratory (hematological, blood chemistry tests). Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator;
* Normal ECG recording on a 12-lead ECG at the screening visit:

  * 120 < PR < 210 ms,
  * QRS < 120 ms,
  * QTcf ≤ 430 ms for male and < 450 ms for female,
  * No sign of any trouble of sinusal automatism,
  * Or considered NCs by investigators;
* Negative prick test at screening visit for the whole study product (extract of Tobacco leaf and NaCL), and positive for histamine;
* French speaking subject;
* Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.
* Subject having signed the informed consent agreement.

Exclusion Criteria:

* Pregnancy and breastfeeding;
* Concomitant participation to another clinical trial;
* Concomitant active infectious diseases;
* Concomitant use of treatment known to interfere with immune response (not including desensitization therapies);
* Uncontrolled diabetes;
* Prior exposure to a nicotine vaccine or to any other vaccine within 30 days before study product administration;
* Concomitant use (and within previous 60 days) of any smoking cessation therapy (including electronic cigarettes and alternative methods such as hypnosis or acupuncture);
* Legal incapacity or physical, psychological or mental status interfering with the subject's ability to sign the informed consent or to terminate the study.
* Subject who would receive more than 4500 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Rate of participants achieving 4-week continuous abstinence | 4-week
  4-weekcontinuous abstinence measured from D15 to D43
Rate of participants achieving 6-month continuous abstinence | 6-month
  6-month continuous abstinence measured from D15 to M6

SECONDARY OUTCOMES:
Rate of participants achieving 12-month continuous abstinence | 12-month
  12-month continuous abstinence measured from D15 to M12
Rate of participants achieving 3-month continuous abstinence | 3-month
  3-month continuous abstinence measured from D15 to M3
Rate of participants achieving 3-month continuous abstinence End of Treatment | 3-month
  continuous abstinence measured during 3-month after end of treatment
Rate of participants achieving 6-month continuous abstinence End of Treatment | 6-month
  continuous abstinence measured during 6-month after end of treatment
Rate of participants achieving 3-month continuous abstinence End of Study | 3-month
  continuous abstinence measured from M9 to M12

CONTACTS AND LOCATIONS:
Overall Officials: Yves Donazzolo, MD, Principal Investigator — Optimed Eurofins
Locations (9):
- France (9):
  - Centre d'Investigation Clinique de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - Eurofins Optimed, Gières
  - Groupe Hospitalier Bretagne Sud, Lorient
  - Centre d'Investigation Clinique de Marseille Nord, Marseille
  - Centre d'Investigation Clinique de Montpellier, Montpellier
  - Centre d'Investigation Clinique de Bordeaux, Pessac
  - Centre d'Investigation Clinique de Poitiers (CIC 1402), Poitiers
  - Centre d'Investigation Clinique de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lafay-Chebassier C, Girodet PO, Laine F, Allain JS, Pickering G, Latreille M, Demina A, Chevassus H, Ingrand I, Tartour E, Benhamouda N, Fraisse ML, Chamitava L, Pletan Y, Balland J, Donazzolo Y, Lafont B. Efficacy and Safety of NFL-101 as a Smoking Cessation Therapy: A Randomized Phase II Clinical Trial CESTO2. Nicotine Tob Res. 2025 Aug 30:ntaf181. doi: 10.1093/ntr/ntaf181. Online ahead of print. PMID 40884488